CLINICAL TRIAL: NCT04199845
Title: Psychophysiological Effects of Lactobacillus Plantarum PS128 in Patients With Major Depressive Disorder :an 8-week Double-blind, Placebo-controlled Trial
Brief Title: 8-week of PS128 RCT in Patients With Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201906056
Record Dates: First submitted 2019-12-10; First posted 2019-12-16 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
Keywords: probiotics; gut permeability; inflammation
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PS128 (Experimental): PS128 will be given twice daily for 8 weeks Active capsule containing 300 mg of probiotics, equivalent to 3 x10^10 CFU of Lactobacillus plantarum PS128.
  Interventions: Dietary Supplement: PS128
- placebo (Placebo Comparator): Placebo containing starch will be given twice daily for 8 weeks.
  Interventions: Dietary Supplement: PS128

INTERVENTIONS:
Dietary Supplement: PS128 — PS128 or placebo will be given twice daily for 8 weeks.

SUMMARY:
Background: Recent studies have suggested that gut-brain axis may be one of the mechanisms of major depression disorder. In animal studies, alteration of gut microbiota can affect animal's depression or anxiety-like behavior, brain neurochemistry and inflammation. In human studies, the composition of gut microbiota is different between patients with MDD and healthy controls. In addition, supplementation of probiotics can improve mood status in community and clinical participants. In preliminary open trial, the investigators found PS-128 can significantly reduce depression severity in patients with MDD. Therefore, the investigators would like to conduct an 8-week randomized, double-blind, placebo controlled trial of PS-128 in patients with MDD.

Aims: This study will be an 8-week randomized, double-blind, placebo-controlled trial to investigate the effects of Lactobacillus plantarum PS128 on psychophysiology in patients with MDD.

Method: This is a two-phase study. In the first phase, the investigators will recruited patients fulfilling the following inclusion criteria: Age 20-65; fulfill Diagnostic and Statistical Manual of Mental Disorders fifth version (DSM-V) criteria of major depressive episode in recent 2 years; Psychotropics including antidepressants, antipsychotics and hypnotics have been kept unchanged for at least 1 months. The exclusion criteria are: comorbid with schizophrenia, bipolar disorder, or other substance use (except tobacco) disorder; having active suicidal or homicidal ideation; known allergy to probiotics; comorbid with diabetes mellitus, irritable bowel syndrome, inflammatory bowl disease, liver cirrhosis, or autoimmune diseases; known active bacterial, fungal, or viral infections in one month; use of antibiotics, steroid, immunosuppressants, probiotics, or synbiotics in the month before collecting blood and fecal samples; pregnant or lactating women; who state to have dietary pattern changed or in diet within previous two months. Those with HAMD-17 >=14 in the first screen will be randomized to PS-128 or placebo, with the ratio of 1:1, in the second phase intervention. In the second phase intervention, the investigators will give eligible patients Lactobacillus plantarum PS128 or placebo for 8 weeks, and compare depression symptoms, gut microbiota, gut permeability, and serum inflammation level before and after intervention.

DETAILED DESCRIPTION:
The eligible patients will be randomly assigned to either active (PS128) or identical-appearing placebo capsule in an 1 : 1 ratio. A research assistant who is blind to the status of participants will conduct the randomization allocation. Recruited patients will be randomized in 1:1 ratio, by a computer-generated allocation sequence with blocks of 4. Patients, caregivers, and investigators will be all masked to the assignment. To ensure the concealment of the randomization assignment, active drug and placebo will be provided by coded containers. At the end of the first year, the investigators will temporarily decode the blinded medication to analyze the preliminary results.

Active capsule containing 300 mg of probiotics, equivalent to 3x10^10 CFU of Lactobacillus plantarum PS128. PS128 and placebo will be manufactured by BENED biomedical and packed by a GMP pharmaceutical manufacture. PS128 or placebo will be provided twice, in the morning and in the afternoon, daily. Because activity and diet may alter composition of gut microbiota, the investigators will ask eligible patients not to change their lifestyle or diet pattern. In addition, though effects of psychotropics on inflammation are still controversial (Baumeister et al. 2016b), medications will be kept unchanged during the intervention period. If kinds of psychotropic were changed because of worsening clinical condition, the patient will be withdrawal from the study. However, if only dose of psychotropics were change, the investigators will record the changes, and the patients will be still kept in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-65
2. fulfill Diagnostic and Statistical Manual of Mental Disorders fifth version (DSM-V) criteria of major depressive episode in recent 2 years
3. Psychotropics including antidepressants, antipsychotics and hypnotics have been kept unchanged for at least one month
4. HAMD-17 >= 14

Exclusion Criteria:

1. Comorbid with schizophrenia, bipolar disorder, or other substance use (except tobacco) disorder.
2. having active suicidal or homicidal ideation
3. known allergy to probiotics
4. comorbid with hypertension, diabetes mellitus, irritable bowel syndrome, inflammatory bowl disease, liver cirrhosis, or autoimmune diseases
5. known active bacterial, fungal, or viral infections in one month.
6. use of antibiotics, steroid, immunosuppressants, probiotics, or synbiotics in the month before collecting blood and fecal samples
7. pregnant or lactating women (by history)
8. who obviously change dietary pattern or in diet within previous month

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Changes of Hamilton Depression Rating Scale- 17 items (HAMD-17) | baseline, week 2, week 4 and week 8.
  HAMD-17 to evaluate the severity of depression

SECONDARY OUTCOMES:
Changes of Depression and Somatic Symptoms Scale (DSSS) | baseline, week 2, week 4 and week 8.
  DSSS to evaluate the severity of depression
Changes of serum zonulin | baseline and week 8
  use serum zonulin and I-FABP to represent gut permeability
Changes of serum IFABP | baseline and week 8
  use serum I-FABP to represent gut permeability
Changes of serum hs-CRP level | baseline and week 8
  inflammation markers
Changes of serum IL-6 level | baseline and week 8
  inflammation markers
Changes of serum IL-10 level | baseline and week 8
  inflammation markers
Changes of serum TNF-alpha level | baseline and week 8
  inflammation markers
Changes of composition of gut microbiota | baseline and week 8
  The investigators will compare the difference of alpha diversity and relative abundance in phylum level, family level, and genus level before and after 8-week PS128 intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hsin Chen, MD, Principal Investigator — TMU-Wan Fang Hospital
Locations (1):
- WanFang Hospital, Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No